CLINICAL TRIAL: NCT04317937
Title: The Effects Of Jaw Sensorimotor System In The Treatment Of Neck Pain And Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Saeed Akhter, principal investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 013
Record Dates: First submitted 2020-03-06; First posted 2020-03-23 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Neck Pain; PHYSIOTHERAPY; JAW
MeSH Terms: conditions — Neck Pain | interventions — Exercise Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaw Movement Group (Experimental): A: Jaw opening-closing movements
  * Active jaw movements
  * Active neck exercises
  B: Isometric strengthening exercises (Same as control group) C: Postural Advice and Home Exercise Program with Dairy (Same as control group)
  Interventions: Other: Jaw opening-closing movements; Other: Exercise Therapy; Other: Supportive Treatment
- Exercise therapy (Active Comparator): A: Active neck exercises Active neck exercises Active jaw movements (Active Jaw movement will not be perform in this group) B: Isometric strengthening exercises C: Postural Advice and Home Exercise Program with Dairy i: Postural Advise ii: Home Exercise Program (unsupervised) iii: Home Dairy
  Frequency and Duration of Treatment Non-specific Chronic Neck Pain (more than 3 months history of pain)
  Initial Assessment (week 1) 60 minutes First treatment session (week1) 40 minutes
  * 3 treatment sessions per week (week- 2) 40 minutes
  * 3 treatment sessions per week (week- 3) 40 minutes
  * 3 treatment sessions per week (week- 4) 40 minutes
  * 3 treatment sessions per week (week- 5) 40 minutes
  * Last treatment session (week 6) 40 minutes
  * Final Assessment (week 6) 60 minutes
  Interventions: Other: Specific Active exercises; Other: Exercise Therapy; Other: Supportive Treatment

INTERVENTIONS:
Other: Jaw opening-closing movements — Jaw opening-closing movements Patient seated on a normal standard comfortable chair with proper back support and feet placed on the floor with no head support.
  Active jaw movements The patient will then perform maximal Jaw opening-closing movements at a pace convenient for his/her for 15 times. Three sets with two minutes rest in between will be ensured.
  Active neck exercises While performing the above movements of jaws, the patient will actively perform active neck exercise (head-neck movements in sagittal plane- Extension- Flexion).
  Head-Neck extension on jaw opening (Mandible moves vertically downward); and then from Head-Neck extension to natural flexion movement on jaw closing (Mandible moves vertically upward).
  Other Names: Jaw movements
  Arms: Jaw Movement Group
Other: Specific Active exercises — Active neck exercises:
  Patient seated on a normal standard comfortable chair with proper back support and feet placed on the floor with no head support.
  Note: For Active neck exercise (flexion and extension movements of neck), firstly the patient will perform maximal Jaw opening-closing movements at a pace convenient for his/her for 5 times in order to observe (eyeball observation) the neck extension and flexion as reference point for each individual.
  Using this reference points, the patient will ask perform below mentioned active neck exercise.
  Active neck exercises: The patient will then perform active neck exercise (flexion and extension of neck) at a pace convenient for his/her for 15 times. Three sets with two minutes rest in between will be ensured.
  Active jaw movement: While performing the above movements of neck, the patient will not perform any jaws movements.
  Other Names: Active neck exercises
  Arms: Exercise therapy
Other: Exercise Therapy — Isometric strengthening exercises For flexion the starting position will be upright head and neck. The patient will be asked to hold this position.
  For extension the starting position will be upright head and neck. The patient will be asked to hold this position.
  For rotation the starting position will be upright head and neck. The patient will be asked to hold this position.
  • In all above movements ( flexion, extension & rotation) following method will be followed: Manual resistance will then be applied by the investigator by placing the hand on the patient's forehead, posterior part of the head and lateral part of the head with 6 second hold. 15 repetitions of this exercise will be performed. Three sets with one minute rest in between will be ensured.
  Other Names: Isometric neck exercises
Other: Supportive Treatment — Postural Advice and Home Exercise Program with Dairy Postural advice and home exercise program. Postural Advise Maintain upright posture while sitting.
  * Avoid prolonged neck bending.
  * Avoid twisting movement of the neck.
  * Use a suitable pillow to maintain cervical spine.
  * Adjust computer screen at eye level.
  * Avoid constant use of mobile or similar device to prevent excessive strain over neck joints and muscles.
  * Carry light and even weight in both hands while shopping and other chores.•Stay hydrated.
  Home Exercise Program (unsupervised) (3 times a day)
  * Forward flexion (Self Resisted), 6 sec hold, number of repetitions 15
  * Right side flexion (Self Resisted ), 6 sec hold, number of repetitions 15
  * Left side flexion (Self Resisted) x 6 sec hold,number of repetitions 15
  * Backward flexion (Self Resisted) x 6 sec hold, number of repetitions 15
  Home Dairy A home dairy will be provided to maintain home exercise program record.
  Other Names: Postural Advice and Home Exercise Program with Dairy

SUMMARY:
The study will be focused on non- specific chronic neck pain patients. The primary objective is to study the effects of jaw sensorimotor system in the treatment of patients with neck pain and dysfunction. It will be randomized controlled trail with the estimated sample size of 80 with both genders. The experimental group will be performed Jaw opening-closing movements with active neck flexion and extension movements and control group will be performed active neck flexion and extension movements. Both groups will be received isometric strengthening exercises, Postural Advice and Home Exercise Program with Dairy. Numeric Pain Rating scale (NPRS), Neck disability Index (NDI), Neck Proprioception tests and Neck muscles endurance test will be used as outcome measures at day 0 and week 6 for treatment effect in both groups. Tables and graphs will used for demographic descriptions and appropriate statistical tests will be applied to establish treatment effect within and between groups.

DETAILED DESCRIPTION:
Study Design : Randomized Controlled Trial

Settings: IPM&R (Institute of Physical Medicine and Rehabilitation). This institute is a part of Dow University of Health Sciences (Karachi-Pakistan).

Duration of study: 18 months after IRB approval

Sample population: Non-specific chronic neck pain

Sample size calculation Using carried out using PASS Version 11 two sample t test with 95% confidence of interval and 80% power of test, mean of NDI (experimental 16.83± 2.3 and 19.13 ± 2.2) calculated sample size is 16 per group which we have increased up to 40 in each group (Experimental & Control) including 8 patients as a dropout rate per group (makes at least 32 patients per group).

Sampling technique: Non probability, purposive sampling technique

Inclusion criteria:

* Both genders
* 18 years to 50 years
* Participants with history neck of more than 3 months with no related conditions
* Non radiating pain to arms
* Diagnosed as Nonspecific Chronic Neck pain by consultants
* NPRS-Numeric Pain Rating Scale score 3 to 8
* NDI- Neck Disability Index : score 5 to 34
* No TMJ pain or dysfunction

Exclusion

* NPRS-Numeric Pain Rating Scale Score 1 & 2 and score 9 & 10 (Score 1 & 2 mild pain and Score 9 & 10 worst pain)
* NDI- Neck Disability Index : Score 0 to 4 (no disability) and score 35 to 50(Complete disability)
* Specific or nonspecific Acute Neck pain (Less than 7 days)
* Neck pain- Specific or nonspecific Sub acute (pain history more than seven days however less than three months)
* Neck pain- Specific Chronic (pain history more than 3 months)
* TMJ Dysfunction
* WAD (Whiplash Associated Disorders)
* Cervical spondylosis
* Rheumatoid arthritis
* Instability of spine
* Facial injury or dental infection
* Any type of infection of body
* Neck or spinal segment fracture
* Spinal tumor or any type of tumor/cancer
* Unexplained headache
* Post cervical spine surgical cases
* Signs and symptoms of Cervical spine stenosis
* Signs and symptoms of disc bulge or herniation of cervical spine
* Radiating neck pain or Radiculopathy of cervical spine
* Cognitive impairment
* Neurological conditions (MS/PD/CVA/MND)
* Application of injection therapy in cervical spine
* Red flags ( Episode of Double vision, Dysarthria, Dysphasia, Drop Attack Dizziness, Double vision, Gait disturbance)

Assessments: After consent filling form, a physiotherapy assessment form will be completed.

Outcome measures (Variables):

i. NPRS ii. NDI iii. Neck Proprioception test iv. Neck Muscles Endurance Test

Treatment assignment (allocation):

In this study, the treatment assignment will be completed using randomization technique.

* In this study, based on inclusion and exclusion criteria, required numbers of sample size participants will recruit first as mentioned earlier using non probability sampling technique.
* Estimated total 80 patients (40 patients per group including dropout rate) (makes at least 32 patients per group) will be selected.
* Total 80 study population will be divided further out in two groups based on gender for giving equal opportunity to participate in this study. 40 male patients (20 for experimental and 20 for control group) and 40 female patients (20 for experimental and 20 for control group) via simple randomization technique using computer generated Microsoft Excel sheet.
* The above mentioned process will be run for male and female parallel or separately depending on the frequency of the patients.

Patients will not be selected in this study based on inclusion criteria, refer to the physiotherapy OPD for assessment and treatment.

Blinding:

* Physiotherapist with minimum two years job experience will be selected and physiotherapist will receive training on how to perform the assessment.
* Treatment blinding will be achieved by asking physiotherapist to complete initial assessment forms with all outcome measures (pre- intervention) to all subjects (referred patients) with non specific chronic neck pain and dysfunction. The physiotherapists will remain unaware about who will be selected as research sample participants including unaware about experimental and control groups.
* At the time of getting consent, patients will be made aware of the relevant details about the research study, however they will remain unaware of their own group allocation.
* The principal investigator alone will administer the treatment.
* The outcome measurements will be taken at day 0 (pre-intervention) and then week 6 outcome measurements (post intervention) will be recorded by physiotherapist.

INTERVENTION: TREATMENT REGIMES FOR EXPERIMENTAL AND CONTROL Experimental group A: Jaw opening-closing movements Active jaw movements Active neck exercises B: Isometric strengthening exercises (Same as control group) C: Postural Advice and Home Exercise Program with Dairy (Same as control group)

Control group:

A: Active neck exercises. B: Isometric strengthening exercises C: Postural Advice and Home Exercise Program with Dairy Postural advice and home exercise program

1. Postural Advise.

   * Maintain upright posture while sitting.
   * Avoid prolonged neck bending.
   * Avoid twisting movement of the neck.
   * Use a suitable pillow to maintain cervical spine.
   * Adjust computer screen at eye level.
   * Avoid constant use of mobile or similar device to prevent excessive strain over neck joints and muscles.
   * Carry light and even weight in both hands while shopping and other chores.
   * Stay hydrated.
2. Home Exercise Program (unsupervised) The following home exercise program will be instructed to all subjects with request to repeat the program 3 times a day.

   * Forward flexion (Self Resisted), 6 sec hold, number of repetitions 15
   * Right side flexion (Self Resisted ), 6 sec hold, number of repetitions 15
   * Left side flexion (Self Resisted) x 6 sec hold,number of repetitions 15
   * Backward flexion (Self Resisted) x 6 sec hold, number of repetitions 15
3. Home Dairy A home dairy will be provided to maintain home exercise program record.

Frequency and Duration of Treatment:

Non-specific Chronic Neck Pain (more than 3 months history of pain) Initial Assessment (week 1) 60 minutes, First treatment session (week1) 40 minutes, 3 treatment sessions per week (week- 2-6 ) 40 minutes, Final Assessment (week 6) 60 minutes.

ETHICAL CONSIDERATIONS

* It will be gained from the Ethical Committee of the University before study
* Written informed consent will be taken from all the patients
* All information and collected data will be kept confidential.
* Participants will remain anonymous throughout the study.
* The Participants will be informed that there are no disadvantages or risks on the procedure of the study.
* Participants will also be informed that they will be free to withdraw at any time during the process of the study.

DATA COLLECTION Data Collection Procedure

* After IRB approval, Data will be collected November 2018 (Subject to approval).
* Collection of data will be initiated once approval of synopsis will be taken.
* Patients will be recruited from IPM&R and consultants will assess and screen patients as indicated and will pass on to physiotherapy department with diagnosed of non specific chronic pain.
* Initial screening proforma will be completed by a physiotherapist based on inclusion and exclusion criteria.
* Non probability sampling technique will be used for recruitment of patients
* A written consent form will be taken from all participants
* Participants will be divided into two groups (Experimental and control groups) as mentioned above.
* Assessment form including outcome measures will be completed on first visit by a trained physiotherapist with experience in the area field of physiotherapy practice at least 2 years.
* The selected outcome measures will be taken on day 0 (pre intervention), and week 6 (post intervention) will be completed by physiotherapist.
* Treatment will be performed for 6 weeks with postural advice and home exercise program with dairy record by principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders

  * 18 years to 50 years
  * Participants with history neck of more than 3 months with no related conditions
  * Non radiating pain to arms
  * Diagnosed as Nonspecific Chronic Neck pain by consultants
  * NPRS-Numeric Pain Rating Scale: score 3 to 8 (Score 3 Ending of mild pain, Score 8 Beginning of worst pain)
  * NDI- Neck Disability Index: score 5 to 34 (5 to 14 Mild disability,15- 24 Moderate disability & 25 to 34 Severity disability)
  * No TMJ pain or dysfunction

Exclusion Criteria:

* • NPRS-Numeric Pain Rating Scale: Score 1 & 2 and score 9 & 10 (Score 1 & 2 mild pain and Score 9 & 10 worst pain)

  * NDI- Neck Disability Index : Score 0 to 4 (no disability) and score 35 to 50(Complete disability)
  * Specific or nonspecific Acute Neck pain (Less than 7 days)
  * Neck pain- Specific or nonspecific Subacute( pain history more than seven days however less than three months)
  * Neck pain- Specific Chronic (pain history more than 3 months)
  * TMJ Dysfunction
  * WAD (Whiplash Associated Disorders)
  * Cervical spondylosis
  * Rheumatoid arthritis
  * Instability of spine
  * Facial injury or dental infection
  * Any type of infection of body
  * Neck or spinal segment fracture
  * Spinal tumor or any type of tumor/cancer
  * Unexplained headache
  * Post cervical spine surgical cases
  * Signs and symptoms of Cervical spine stenosis
  * Signs and symptoms of disc bulge or herniation of cervical spine
  * Radiating neck pain or Radiculopathy of cervical spine
  * Cognitive impairment
  * Neurological conditions (MS/PD/CVA/MND)
  * Application of injection therapy in cervical spine
  * Red flags ( Episode of Double vision, Dysarthria, Dysphasia, Drop Attack, Dizziness, Double vision, Gait disturbance)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating scale (NPRS) | Week 6
  Assessing the change in pain level:
  The subject will be graphically or verbally portrayed a simple depiction consisting of a horizontal bar with labels ranging from '0' to '10' (a total of 11 integers)to rate his pain intensity.'0' would be considered as 'no pain'and '10' would indicate worst pain imaginable, whereas values 1 to 3 would indicate mild pain; 4 to 6 as moderate pain and 7 to 10 would indicate severe pain. NPRS has shown to have good sensitivity and it yields data that are best suited for statistical analysis.
Neck disability Index (NDI) | Week 6
  Assessing the change in neck disability level:
  The Neck Disability Scale is a reliable outcome measure to assess the treatment effectiveness for neck disability. It consists of 10 components.
Neck Proprioception test | Week 6
  Assessing the change in neck preconception error:
  The concept adopted from Hallgren and co workers and it will be used as research instrument on baseline and final visits to find out any proprioceptive errors.
  A Neutral Reference Point (NRP) will be used and asking patient to perform cervical spine range of motion (rotation, flexion and extension). Then measures any overshoot or undershoot of movement with regard to NRP/Starting position using a cervical spine range of motion device.
Neck muscles endurance test | Week 6
  Assessing the change in neck muscle endurance level:
  Neck flexor muscle endurance test will be used to measure neck endurance in this study. It is a simple test and easy to apply. It is reliable test and achieved interrater reliability at moderate level among neck pain population.
  Cervical extensor endurance test is a simple test for measurement neck extensor muscles endurance. It has good inter-rater reliability Kappa =0.800, Kappa SE= 0.109, 95% CL) and easy to administer. Losing of chin tuck position from neutral position of cervical spine is indicating of global weakness of neck muscles (weakness of superficial and deep neck extensor muscles) whist increasing of chin length with neck extension indicates a over activity of superficial extensor muscles and weakness of deep extensor muscles of cervical spine.

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Akhter, MS, Principal Investigator — University of Lahore
Locations (1):
- Insititute of Physical Medicine & Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Eriksson PO, Haggman-Henrikson B, Nordh E, Zafar H. Co-ordinated mandibular and head-neck movements during rhythmic jaw activities in man. J Dent Res. 2000 Jun;79(6):1378-84. doi: 10.1177/00220345000790060501. PMID 10890716
- [Background] Loeser JD, Treede RD. The Kyoto protocol of IASP Basic Pain Terminology. Pain. 2008 Jul 31;137(3):473-477. doi: 10.1016/j.pain.2008.04.025. Epub 2008 Jun 25. No abstract available. PMID 18583048
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Sihawong R, Janwantanakul P, Sitthipornvorakul E, Pensri P. Exercise therapy for office workers with nonspecific neck pain: a systematic review. J Manipulative Physiol Ther. 2011 Jan;34(1):62-71. doi: 10.1016/j.jmpt.2010.11.005. PMID 21237409
- [Background] Genebra CVDS, Maciel NM, Bento TPF, Simeao SFAP, Vitta A. Prevalence and factors associated with neck pain: a population-based study. Braz J Phys Ther. 2017 Jul-Aug;21(4):274-280. doi: 10.1016/j.bjpt.2017.05.005. Epub 2017 May 20. PMID 28602744
- [Background] Malchaire JB, Roquelaure Y, Cock N, Piette A, Vergracht S, Chiron H. Musculoskeletal complaints, functional capacity, personality and psychosocial factors. Int Arch Occup Environ Health. 2001 Oct;74(8):549-57. doi: 10.1007/s004200100264. PMID 11768043
- [Background] Cimmino MA, Ferrone C, Cutolo M. Epidemiology of chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):173-83. doi: 10.1016/j.berh.2010.01.012. PMID 22094194
- [Background] Vasseljen O, Woodhouse A, Bjorngaard JH, Leivseth L. Natural course of acute neck and low back pain in the general population: the HUNT study. Pain. 2013 Aug;154(8):1237-44. doi: 10.1016/j.pain.2013.03.032. Epub 2013 Apr 2. PMID 23664654
- [Background] Vos CJ, Verhagen AP, Passchier J, Koes BW. Clinical course and prognostic factors in acute neck pain: an inception cohort study in general practice. Pain Med. 2008 Jul-Aug;9(5):572-80. doi: 10.1111/j.1526-4637.2008.00456.x. Epub 2008 Jun 28. PMID 18565009
- [Background] Pernold G, Mortimer M, Wiktorin C, Tornqvist EW, Vingard E; Musculoskeletal Intervention Center-Norrtalje Study Group. Neck/shoulder disorders in a general population. Natural course and influence of physical exercise: a 5-year follow-up. Spine (Phila Pa 1976). 2005 Jul 1;30(13):E363-8. doi: 10.1097/01.brs.0000167819.82642.f7. PMID 15990653
- [Background] Christensen JO, Knardahl S. Time-course of occupational psychological and social factors as predictors of new-onset and persistent neck pain: a three-wave prospective study over 4 years. Pain. 2014 Jul;155(7):1262-1271. doi: 10.1016/j.pain.2014.03.021. Epub 2014 Apr 2. PMID 24704365
- [Background] Carstensen TB. The influence of psychosocial factors on recovery following acute whiplash trauma. Dan Med J. 2012 Dec;59(12):B4560. PMID 23290295
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Sharmila B. Isometric muscle energy technique and non-specific neck pain in secondary school teachers-Results of an experimental study.Indian J Physiother Occup Ther. 2014;8(2):58.
- [Background] Dubner R, Ren K, Sessle BJ. Sensory mechanisms of orofacial pain: Intreatment of TMDs: Bridging the Gap. Pain. 2013;154:511-14.
- [Background] Avivi-Arber L, Martin R, Lee JC, Sessle BJ. Face sensorimotor cortex and its neuroplasticity related to orofacial sensorimotor functions. Arch Oral Biol. 2011 Dec;56(12):1440-65. doi: 10.1016/j.archoralbio.2011.04.005. Epub 2011 May 8. PMID 21550585
- [Background] McLoon LK, Andrade F. Craniofacial muscles: A new framework for understanding the effector side of craniofacial muscle control. Springer Science & Business Media. 2013:111-30.
- [Background] Leston JM. [Functional anatomy of the trigeminal nerve]. Neurochirurgie. 2009 Apr;55(2):99-112. doi: 10.1016/j.neuchi.2009.01.001. Epub 2009 Mar 19. French. PMID 19303117
- [Background] De Laat A, Meuleman H, Stevens A, Verbeke G. Correlation between cervical spine and temporomandibular disorders. Clin Oral Investig. 1998 Jun;2(2):54-7. doi: 10.1007/s007840050045. PMID 15490776
- [Background] de Wijer A, Steenks MH, de Leeuw JR, Bosman F, Helders PJ. Symptoms of the cervical spine in temporomandibular and cervical spine disorders. J Oral Rehabil. 1996 Nov;23(11):742-50. doi: 10.1046/j.1365-2842.1996.d01-187.x. PMID 8953478
- [Background] Piovesan EJ, Kowacs PA, Oshinsky ML. Convergence of cervical and trigeminal sensory afferents. Curr Pain Headache Rep. 2003 Oct;7(5):377-83. doi: 10.1007/s11916-003-0037-x. PMID 12946291
- [Background] Binder AI. Cervical spondylosis and neck pain. BMJ. 2007 Mar 10;334(7592):527-31. doi: 10.1136/bmj.39127.608299.80. No abstract available. PMID 17347239
- [Background] Bruflat AK, Balter JE, McGuire D, Fethke NB, Maluf KS. Stress management as an adjunct to physical therapy for chronic neck pain. Phys Ther. 2012 Oct;92(10):1348-59. doi: 10.2522/ptj.20110489. Epub 2012 Jun 14. PMID 22700538
- [Background] Cote P, van der Velde G, Cassidy JD, Carroll LJ, Hogg-Johnson S, Holm LW, Carragee EJ, Haldeman S, Nordin M, Hurwitz EL, Guzman J, Peloso PM. The burden and determinants of neck pain in workers: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S70-86. doi: 10.1016/j.jmpt.2008.11.012. PMID 19251078
- [Background] Chiu TW, Leung SL, Lam KW. Neck pain in Hong Kong: a telephone survey on consequences and health service utilisation. Hong Kong Med J. 2012 Aug;18 Suppl 3:13-5. No abstract available. PMID 22865216
- [Background] Skillgate E, Magnusson C, Lundberg M, Hallqvist J. The age- and sex-specific occurrence of bothersome neck pain in the general population--results from the Stockholm public health cohort. BMC Musculoskelet Disord. 2012 Sep 24;13:185. doi: 10.1186/1471-2474-13-185. PMID 23006655
- [Background] Falco FJ, Manchikanti L, Datta S, Wargo BW, Geffert S, Bryce DA, Atluri S, Singh V, Benyamin RM, Sehgal N, Ward SP, Helm S 2nd, Gupta S, Boswell MV. Systematic review of the therapeutic effectiveness of cervical facet joint interventions: an update. Pain Physician. 2012 Nov-Dec;15(6):E839-68. PMID 23159978
- [Background] Lauche R, Cramer H, Langhorst J, Dobos G, Gerdle B. Neck pain intensity does not predict pressure pain hyperalgesia: re-analysis of seven randomized controlled trials. J Rehabil Med. 2014 Jun;46(6):553-60. doi: 10.2340/16501977-1815. PMID 24715237
- [Background] Martel J, Dugas C, Dubois JD, Descarreaux M. A randomised controlled trial of preventive spinal manipulation with and without a home exercise program for patients with chronic neck pain. BMC Musculoskelet Disord. 2011 Feb 8;12:41. doi: 10.1186/1471-2474-12-41. PMID 21303529
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Sowmya MV. Isometric neck exercises versus dynamic neck exercises in chronic neck pain. 2014;3(2):32-43
- [Background] Pillastrini P, de Lima E Sa Resende F, Banchelli F, Burioli A, Di Ciaccio E, Guccione AA, Villafane JH, Vanti C. Effectiveness of Global Postural Re-education in Patients With Chronic Nonspecific Neck Pain: Randomized Controlled Trial. Phys Ther. 2016 Sep;96(9):1408-16. doi: 10.2522/ptj.20150501. Epub 2016 Mar 24. PMID 27013576
- [Background] Beltran-Alacreu H, Lopez-de-Uralde-Villanueva I, Fernandez-Carnero J, La Touche R. Manual Therapy, Therapeutic Patient Education, and Therapeutic Exercise, an Effective Multimodal Treatment of Nonspecific Chronic Neck Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2015 Oct;94(10 Suppl 1):887-97. doi: 10.1097/PHM.0000000000000293. PMID 25888653
- [Background] Pöntinen PJ. Reliability, validity, reproducibility of algometry in diagnosis of active and latent tender spots and trigger points. J Musculoskelet Pain. 1998;6(1):61-71.
- [Background] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Background] Young BA, Walker MJ, Strunce JB, Boyles RE, Whitman JM, Childs JD. Responsiveness of the Neck Disability Index in patients with mechanical neck disorders. Spine J. 2009 Oct;9(10):802-8. doi: 10.1016/j.spinee.2009.06.002. Epub 2009 Jul 25. PMID 19632904
- [Background] Salo P, Ylinen J, Kautiainen H, Arkela-Kautiainen M, Hakkinen A. Reliability and validity of the finnish version of the neck disability index and the modified neck pain and disability scale. Spine (Phila Pa 1976). 2010 Mar 1;35(5):552-6. doi: 10.1097/BRS.0b013e3181b327ff. PMID 20147882
- [Background] Hallgren RC, Andary MT. Undershooting of a neutral reference position by asymptomatic subjects after cervical motion in the sagittal plane. J Manipulative Physiol Ther. 2008 Sep;31(7):547-52. doi: 10.1016/j.jmpt.2008.08.011. PMID 18804006
- [Background] Rheault W, Albright B, Beyers C, Franta M, Johnson A, Skowronek M, Dougherty J. Intertester reliability of the cervical range of motion device. J Orthop Sports Phys Ther. 1992;15(3):147-50. doi: 10.2519/jospt.1992.15.3.147. PMID 18796788
- [Background] Youdas JW, Carey JR, Garrett TR. Reliability of measurements of cervical spine range of motion--comparison of three methods. Phys Ther. 1991 Feb;71(2):98-104; discussion 105-6. doi: 10.1093/ptj/71.2.98. PMID 1989013
- [Background] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Background] Sebastian D, Chovvath R, Malladi R. Cervical extensor endurance test: a reliability study. J Bodyw Mov Ther. 2015 Apr;19(2):213-6. doi: 10.1016/j.jbmt.2014.04.014. Epub 2014 Apr 18. PMID 25892374
- [Background] Akhter S, Khan M, Ali SS, Soomro RR. Role of manual therapy with exercise regime versus exercise regime alone in the management of non-specific chronic neck pain. Pak J Pharm Sci. 2014 Nov;27(6 Suppl):2125-8. PMID 25410083
- [Background] Zar JH. Biostatistical Analysis. 4th ed. New Jersey: Pearson; 2010.
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Hafeez A. Urdu version of the neck disability index: a reliability and validity study. BMC Musculoskelet Disord. 2017 Apr 8;18(1):149. doi: 10.1186/s12891-017-1469-5. PMID 28388888
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732